CLINICAL TRIAL: NCT01060228
Title: An Open-Label, Drug-Drug Interaction Study Between Steady-State Valproic Acid and Single-Dose Paliperidone Extended-Release in Healthy Men
Brief Title: A Drug Interaction Study of Valproic Acid and Single-dose Paliperidone Extended-Release (ER) in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CR015802; R076477BIM1003
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Schizophrenia; Epilepsy
Keywords: Paliperidone ER; INVEGA; Divalproex sodium; Depakote ER; Pharmacokinetics; Valproic Acid; Human Experimentation
MeSH Terms: conditions — Schizophrenia; Epilepsy | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Other): paliperidone ER 1 tablet of 500 mg once daily on Day 1 and Day 15
  Interventions: Drug: paliperidone ER
- 002 (Other): divalproex sodium ER 2 tablets of 500 mg once daily from Days 5 through 18
  Interventions: Drug: divalproex sodium ER

INTERVENTIONS:
Drug: paliperidone ER — 1 tablet of 500 mg once daily on Day 1 and Day 15
  Arms: 001
Drug: divalproex sodium ER — 2 tablets of 500 mg once daily from Days 5 through 18
  Arms: 002

SUMMARY:
The purpose of this study is to evaluate the effect of valproic acid (VPA) on the pharmacokinetics (blood levels) of a single oral dose of an extended-release formulation of paliperidone in healthy male volunteers.

DETAILED DESCRIPTION:
This is an open-label (patient will know the identity of the study drug they are taking) study in healthy volunteers (only healthy men will be asked to participate in the study). The primary purpose of the study is to determine how paliperidone (a schizophrenia medication) and divalproex sodium (an epilepsy medication also referred to as valproic acid [VPA]) interact with each other to affect the absorption, distribution, metabolism, and elimination by the body. Other purposes of the study are to learn about the safety of the two study drugs when taken together and to learn how healthy volunteers tolerate the two drugs when taken together. Approximately 24 healthy men (referred to as healthy volunteers) will take part in the study. The study will last about 40 days and will consist of a screening period beginning up to 21 days before the first study drug administration followed by an open label treatment period that will last approximately 20 days (Day -1 through Day 19). The purpose of the screening visit is to see if healthy volunteers meet all of the requirements to participate in the study. During the screening period which may require more than one visit to the study clinic, the following procedures will be performed: 1) signed informed consent will be obtained from healthy volunteers to document that they agree to participate in the study, 2) medical history and demographic information including age, date of birth, sex, race, etc will be collected, 3) a physical examination will be performed, 4) vital signs (pulse rate, blood pressure, and temperature) will be measured, 5) a blood sample will be collected for routine laboratory tests as well as to test for hepatitis B, hepatitis C, and human immunodeficiency virus (HIV), and 6) a urine sample will be collected for routine laboratory testing including testing for drugs of abuse and alcohol. Healthy volunteers who meet the entry criteria for enrollment at screening will be asked to check in to the study clinic the evening before the first administration of study drug (Day -1) and will stay overnight in the clinic until Day 19. During the 20 days at the study clinic, healthy volunteers will be asked to refrain from the consumption of food or beverages containing alcohol, grapefruit juice, Seville oranges, or quinine (such as tonic water), use of any caffeine/xanthine-containing products (coffee, tea, chocolate, cola, other soda with caffeine), and food containing poppy seeds. Healthy volunteers will also be asked to refrain from jogging, strenuous exercise of all types, and sunbathing while confined to the study center and for 48 hours before admission to the study center. Healthy volunteers will be provided with standard meals during the 20 days of confinement at the study center and may smoke throughout the study with a limit of 10 cigarettes or 2 cigars, or 2 pipes of tobacco per day. If a healthy volunteer has an illness with a fever within 2 days of a scheduled dose of study drug, the dose of study drug will be postponed until their body temperature is normal for at least 72 hours (3 days). All healthy volunteers will take each study drug orally (by mouth) in the following order on the days specified: 1 extended release (ER) tablet of 12 mg paliperidone on Day 1 followed by two 500-mg ER tablets of divalproex sodium once daily from Day 5 to 18, and 1 tablet of 12 mg paliperidone ER on Day 15. Paliperidone ER tablets will be taken by healthy volunteers after an overnight fast (having nothing to eat or drink except water) of at least 10 hours. Divalproex sodium ER tablets can be taken at any time between 1 hour before and 1 hour after a meal (except for Days 14 and 15); the morning dose on Days 14 and 15 will be administered after a 10 hour fast. All study drug tablets will be swallowed whole with a glass of water (tablets must not chewed, divided, dissolved, or crushed). The shells of the paliperidone ER tablets are non-disintegrating and may leave the body intact. Therefore, healthy volunteers may see the shells of the tablets in their stools but there is no reason for alarm. During the study, healthy volunteers will have blood samples taken from a vein in their arm using a needle. Each blood sample will consist of approximately 1 teaspoonful of blood. Over the course of the study a total of 53 blood samples will be collected which is about a total of 9 ounces or just a little over a cup of blood. The blood samples will be used to evaluate the primary outcome measure in the study which is the pharmacokinetics (blood levels) of a single dose of orally administered paliperidone ER before and during the administration of VPA at steady-state (steady state is achieved when the rate of drug absorption equals that of the drug elimination and drug concentrations in blood are stable). Healthy volunteers will also be monitored for safety throughout the study. Safety assessments include monitoring of adverse events (side effects) and findings from clinical laboratory tests (including hematology, serum chemistry, and urinalysis), 12-lead electrocardiograms (ECGs) (ECGs are used to trace the electrical activity of the heart), vital signs measurements, and physical examinations. A review of concomitant medications/therapies taken by healthy volunteers during the study will also be performed. Healthy volunteers will complete the study after the final blood sample is collected on Day 19. Before leaving the study center, end of study procedures performed will include a physical examination, vital signs measurements, routine clinical laboratory tests, and an ECG. All healthy volunteers will receive a single oral (by mouth) dose of one 12 mg paliperidone extended release (ER) tablet on Day 1 followed by two 500-mg divalproex sodium ER tablets (each tablet equivalent to 500 mg of valproic acid) for oral administration once daily from Day 5 to 18 and a single oral dose of one 12 mg paliperidone ER tablet on Day 15. All drugs will be swallowed with 240 mL of noncarbonated water and must be swallowed whole, not chewed, divided, dissolved, or crushed.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained indicating an understanding of the purpose of and procedures required for the study and willingness to participate in the study
* Agree to use an adequate contraception method as deemed appropriate by the study physician (for example, vasectomy, double-barrier, partner using effective contraception) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Have a body mass index (BMI, weight [kg]/height2 [m]2) between 18 and 30 kg/m2 (inclusive) and body weight not less than 50 kg
* Have a systolic blood pressure between 90 and 140 mm Hg and a diastolic blood pressure between 50 and 90 mm Hg
* Habitually smokes no more than 10 cigarettes, or 2 cigars, or 2 pipes of tobacco per day for at least 6 months before first study drug administration

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) drug or alcohol abuse within the past 5 years, cancer with exception of basal cell carcinoma, epilepsy, suspected urea cycle disorder, any severe pre-existing gastrointestinal narrowing or malabsorption problems, cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the study physician considers should exclude the healthy volunteer or that could interfere with the interpretation of the study results
* Known allergy or intolerance to study drugs including paliperidone, valproic acid (VPA), sodium valproate, or divalproex sodium or any of the excipients (inactive substances) of the drugs (such as lactose)
* Donated blood or blood products or had substantial loss of blood (more than 500 mL) within 3 months before the first administration of study drug or intention to donate blood or blood products during the study or within 1 month after the completion of the study
* Unable to swallow solid, oral dosage forms whole with the aid of water (participants may not chew, divide, dissolve, or crush the study drugs)
* Preplanned surgery or procedures that would interfere with the conduct of the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-01; Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics of a single dose of orally administered paliperidone ER before and during the administration of VPA at steady-state | Blood samples taken within 2 hours before dosing on Day 1, and during 96 hours after dosing on Day 15 with paliperidone ER

SECONDARY OUTCOMES:
To determine the effect of a single dose of paliperidone ER on steady-state VPA plasma concentrations | Predose on Days 12 to 16, and 19
To evaluate safety and tolerability of the 12-mg tablet of paliperidone ER administered with and without divalproex sodium ER | Day -1 through the last study assessment on Day 19.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: An Open-Label, Drug-Drug Interaction Study between Steady-State Valproic Acid and Single-Dose Paliperidone Extended-Release in Healthy Men — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=799&filename=CR015802_CSR.pdf